CLINICAL TRIAL: NCT03981588
Title: CARDIOTOXICITY IN THE ELDERLY
Acronym: CARTIER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: AORTICA Group (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Principal Investigator, Pedro L Sanchez, Head of the Cardiology Department, AORTICA Group
Other Study IDs: PIE14/00066
Record Dates: First submitted 2019-06-06; First posted 2019-06-11 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2019-06

CONDITIONS: Cardiotoxicity; Elderly; Cardiac Magnetic Resonance
MeSH Terms: conditions — Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Imaging studies — Patients will undergo different imaging and clinical follow-up procedures to run out cardiotoxicity

SUMMARY:
CARTIER (Cardiotoxicity in the elderly) is a prospective cohort study of newly diagnosed elderly cancer patients equal or greater than 65 years of age conduced in one tertiary center (Hospital Universitario de Salamanca at Spain. The study is academically funded in its integrity by The Instituto de Salud Carlos III (Spanish Ministry of Science, Innovation and Universities). The investigators of the study are the only responsible for the study design, data collection, and data interpretation. All study participants provide written informed consent. All enrolled patients will undergo serial surveys, 6-minutes walking test (6MWT), electrocardiogram, echocardiogram, blood samples, CMR, physical examinations and multidisciplinary clinical evaluations; before each chemotherapy cycle and at 3, 6, 9 and 12 months, 3 years and 5 years after finalization of chemotherapy, except for MRI that will be performed before 1st, 3rd, 5th cycles and at 3, 6, 9,12 months, 3 years and 5 years after chemotherapy ending

DETAILED DESCRIPTION:
Surveys completion and examinations will be obtained at the same day: within 72 hours before each cycle of treatment or at 3, 6, 9, 12 months, 3 years and 5 years' follow-up after ending the whole antitumoral course of treatment. A fully dedicated research nurse will play a vital role in ensuring that the study run smoothly and that all participants will be safe and fully informed. Questionnaires completion and quality of life assessment will initially be performed followed by the 6MWT. Participants blood pressure measurement, electrocardiogram and echocardiogram will be then taken >30 minutes after finishing the walking test. Blood sample extraction will be performed after echocardiography to finalize with cardiac magnetic resonance. A complete medical history, physical examination and evaluation of these examinations for each participant will be performed by a cardiologist at the cardio-oncology unit, where prevention and treatment protocols for cardiotoxicity will be applied and discussed in a multidisciplinary way with referral oncologists and hematologists before every cycle of treatment and after course of antitumoral ending follow-up.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed cancer initiating antisudoral treatment
* capability to sign the informed consent
* capability to realize 6 minutes walking test

Exclusion Criteria:

* previous chemotherapy
* contraindications to undergo cardiac magnetic resonance (CMR)
* enrollment in onco-hematologist current clinical-trials
* clinical situation making difficult the realization of the proposed examinations or the course of chemotherapy.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with newly diagnosed cancer initiating antisudoral treatment
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiotoxicity | 5 years
  53% as the lower limit of ejection fraction regardless of gender

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario de Salamanca, Salamanca
  - Pedro Dorado, Salamanca

IPD SHARING:
Plan to Share IPD: Undecided